CLINICAL TRIAL: NCT00058253
Title: A Phase I Study of 17-N-Allylamino-17-Demethoxy Geldanamycin (17-AAG, NSC# 330507) in Combination With Docetaxel in Patients With Advanced Solid Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01436; NCI-2012-01436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5878; CDR0000287199; MSKCC-03006; 03-006 (Other: Memorial Sloan-Kettering Cancer Center); 5878 (Other: CTEP); P30CA008748 (NIH); U01CA069856 (NIH)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Prostate Cancer; Stage IV Prostate Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tanespimycin; Docetaxel

ARMS (2):
- Group I (Experimental): Patients receive docetaxel IV over 1 hour and 17-AAG IV over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tanespimycin; Drug: docetaxel
- Group II (Experimental): Patients receive docetaxel IV over 30 minutes and 17-AAG as in group 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tanespimycin; Drug: docetaxel

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT

SUMMARY:
This phase I trial is studying the side effects and best dose of combination chemotherapy in treating patients with metastatic or unresectable solid tumors. Drugs used in chemotherapy, such as docetaxel and 17-N-allylamino-17-demethoxygeldanamycin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) administered with docetaxel in patients with progressive metastatic prostate cancer or other progressive metastatic or unresectable solid tumors.

II. Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose-escalation study of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG). Patients are assigned to 1 of 2 treatment groups.

Group 1: Patients receive docetaxel IV over 1 hour and 17-AAG IV over 1-2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Group 2: Patients receive docetaxel IV over 30 minutes and 17-AAG as in group 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients per group receive escalating doses of 17-AAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 20 additional patients (10 per group) are treated at the MTD.

Patients are followed every 2-3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or unresectable malignancy for which standard curative or palliative therapy does not exist or is no longer effective
* Progressive disease manifested by the following parameters

  * For prostate cancer:

    * Must have castrate, metastatic disease defined by disease progression after surgical castration or treatment with a gonadotropin-releasing hormone (GnRH) analog (testosterone level less than 50 ng/mL)

      * Patients who have not undergone surgical orchiectomy should continue on medical therapies to maintain castrate levels of testosterone
    * Progressive metastatic disease on imaging studies (bone scan, CT scan, or MRI) OR metastatic disease and a rising prostate-specific antigen (PSA)
    * Biochemical progression indicated by at least 3 rising PSA values (obtained at least 1 week apart) from a baseline OR 2 rising PSA values (more than 1 month apart), where the percentage increase over the range of values is at least 25%
    * Patients who have received an antiandrogen as part of first-line hormonal therapy must have shown progression of disease off of the antiandrogen prior to study enrollment
  * For other solid tumors:

    * Development of new lesions or an increase in pre-existing lesions by bone scintigraphy, CT scan, MRI, positron emission tomography, or physical examination
    * Patients whose sole criterion for progression is an increase in a biochemical marker (e.g., carcinoembryonic antigen or CA 15-3) or an increase in symptoms are not eligible
* Patients with metastatic disease must not be progressing to the extent as to require palliative treatment within 4 weeks of study entry
* No active brain metastases
* Performance status - Karnofsky 70-100%
* More than 6 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT < 1.5 times ULN
* PT ≤ 1.1 times ULN
* Creatinine no greater than 1.4 mg/dL or within ULN
* Creatinine clearance greater than 55 mL/min
* No prior history of pulmonary toxicity after receiving anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone hydrochloride, bleomycin, or carmustine)
* No dyspnea ≥ grade 2 at rest on room air
* No requirement for supplementary oxygen therapy or oxygen saturations ≤ 88%
* No clinically significant pulmonary comorbidities that require medication (e.g., severe chronic obstructive pulmonary disease that could predispose patient to pulmonary toxicity)
* QTc ≤ 450 msec for male patients (470 for female patients)
* LVEF > 40% by echocardiogram or MUGA
* Echocardiogram or MUGA required for patients with any of the following:

  * Myocardial infarction > 1 year ago
  * NYHA class I or II CHF
  * Atrial fibrillation
  * Right or left bundle branch block by EKG
* No history of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No myocardial infarction within the past year
* No active ischemic heart disease within the past year
* No New York Heart Association (NYHA) class III or IV congestive heart failure (CHF)
* No poorly controlled angina
* No uncontrolled dysrhythmia
* No congenital long QT syndrome
* No left bundle branch block
* No other significant cardiac disease
* No prior history of cardiac toxicity after receiving anthracyclines such as doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone hydrochloride, bleomycin, or carmustine
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of severe hypersensitivity reaction to paclitaxel, docetaxel, or polysorbate 80
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No grade 2 or greater symptomatic peripheral neuropathy
* No allergy to eggs or egg products
* No other concurrent uncontrolled illness
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy to sole measurable lesion
* No prior mantle-field radiotherapy
* See Disease Characteristics
* No concurrent surgery for sole measurable lesion
* Recovered from prior therapy
* At least 1 week since prior ketoconazole and recovered
* At least 4 weeks since prior investigational anticancer therapeutic drugs
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent medications that prolong QTc interval
* No concurrent medication used to control arrhythmias

  * Calcium blockers and beta blockers allowed
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies (investigational or commercial)
* No concurrent CYP3A4 inhibitors, including any of the following:

  * Fluconazole
  * Itraconazole
  * Ketoconazole
  * Macrolide antibiotics (azithromycin, clarithromycin, erythromycin, or troleandomycin)
  * Nifedipine
  * Verapamil
  * Diltiazem
  * Cyclosporine
  * Grapefruit juice
* No concurrent CYP3A4 inducers, including any of the following:

  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * Rifampin
* No concurrent herbal extracts or tinctures with CYP3A4 inhibitory activity, including any of the following:

  * Hydrastis canadensis (goldenseal)
  * Hypericum perforatum (St. John's wort)
  * Uncaria tomentosa (cat's claw)
  * Echinacea angustifolia roots
  * Trifolium pratense (wild cherry)
  * Matricaria chamomilla (chamomile)
  * Glycyrrhiza glabra (licorice)
  * Dillapiol
  * Hypericin
  * Naringenin
* Concurrent CYP3A4 substrates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-02; Primary Completion 2008-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose determined by dose-limiting toxicities assessed using the NCI Common Toxicity Criteria (CTC) version 2.0 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: David Solit, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States